CLINICAL TRIAL: NCT05549908
Title: Randomized, Blind, Phase III Clinical Trial to Evaluate the Immunogenicity and Safety of Freeze-dried Human Rabies Vaccine (Vero Cell) Inoculated in 4-dose Program (2-1-1)
Brief Title: Vaccine Prevention of Rabies Adopts 4-shot Immunization Method
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun Zhuoyi Biological Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZY201905001
Record Dates: First submitted 2022-09-14; First posted 2022-09-22 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-02

CONDITIONS: Rabies Human; Antibody Titer
MeSH Terms: interventions — Rabies Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental 4 doses (Experimental): Inoculate experimental vaccine according to 2-1-1 immunization procedure
  Interventions: Biological: rabies vaccine
- Experimental 5 doses (Experimental): Inoculate experimental vaccine according to 1-1-1-1-1 immunization procedure
  Interventions: Biological: rabies vaccine
- SPEEDA® 4 doses (Active Comparator): Inoculate SPEEDA® according to 2-1-1 immunization procedure
  Interventions: Biological: rabies vaccine

INTERVENTIONS:
Biological: rabies vaccine — The subjects were vaccinated with rabies vaccines with different immunization procedures, and the safety and immunogenicity were compared

SUMMARY:
A phase III clinical trial to evaluate the immunogenicity and safety of freeze-dried human rabies vaccine (Vero cell) developed by Changchun Zhuoyi Biological Co., Ltd. inoculated in a 4-dose procedure (2-1-1)

DETAILED DESCRIPTION:
It is to prove that the freeze-dried human rabies vaccine (Vero cell) in the population aged 10-60 years, the four dose vaccination program is not inferior to the five dose vaccination program, and the safty、antibody positive conversion rate and geometric mean concentration of the four dose group of the test vaccine are not inferior to the five dose program group 14 days after the first dose vaccination.

To compare the immunogenicity of people aged 10-60 years old who were vaccinated 6 and 12 months after the whole vaccination, so as to evaluate the antibody positive rate and GMT 6 and 12 months after the test vaccine was vaccinated.

ELIGIBILITY:
Inclusion Criteria:

* The age is 10-60 years old;
* Underarm temperature ≤ 37.0 ℃.

Exclusion Criteria:

* Have a history of rabies vaccine immunization or use of rabies virus passive immunization agents；
* Has been diagnosed with congenital or acquired immunodeficiency disease；
* Pregnancy (including positive urine pregnancy test) or lactation, planned pregnancy preparation within 2 months.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1800 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Antibody positive conversion rate of experimental groups | 3 months
  - Compare the Antibody positive conversion rate between two experimental groups 14 days after the first dose of inoculation.
Antibody positive conversion rate of 4 doses groups | 3 months
  -Compare the Antibody positive conversion rate between the SPEEDA 4 doses group and experimental 4 doses group 14 days after the first dose of inoculation.
Compare the GMT between two experimental groups | 3 months
  - Compare the GMT between two experimental groups 14 days after the first dose of inoculation.
Geometric Mean Titer (GMT) of 4 doses groups | 3 months
  - Compare the GMT between the SPEEDA 4 doses group and the experimental 4 doses group 14 days after the first dose inoculation.
Safety within 30 minutes | 3 months
  - Incidence rate of any local and systemic adverse events (AE) within 30 minutes after each dose of inoculation;
Safety within 0-7 days | 3 months
  - Incidence rate of collected AE within 0-7 days after each dose of inoculation;
Safety within 6 months | 9months
  - Incidence rate of all serious adverse events (SAE) within 6 months from the first dose of inoculation to the full course of inoculation.

SECONDARY OUTCOMES:
Antibody test of 7 days. | 3 months
  - Antibody test 7 days after the first dose of inoculation.
Antibody test after whole vaccination. | 3 months
  - Antibody test 14days after the whole vaccination.
Persistent observation within 12 months | 16 months
  - Antibody test in different points within 12 months after the whole vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Li Miao, Dr, Study Director — Changchun Zhuoyi Biological Co., Ltd
Locations (1):
- Changchun Zhuoyi Biological Co., Ltd, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
all results.
Supporting Information: Study Protocol
Time Frame: before December 2023.
Access Criteria: public for all.

REFERENCES:
- [Derived] Jin F, Zhu L, Wang Y, Qin G, Tian Y, Xie Y, Jin H, Zhang Y, Wang L, Li J, Wu Z, Sheng Y, Shi L, Yang G, Zhao Z, Chen L, Chen P, Jiang Z, Yu J, Gao Z, Li Q, Wu X, Miao L. Randomized, blind, controlled phase III clinical trial: Assessing the immunogenicity and safety of freeze-dried human rabies vaccine (vero cell) with a 4-dose regimen (2-1-1) in a 10-60 year-old demographic. Vaccine. 2024 Oct 3;42(23):126059. doi: 10.1016/j.vaccine.2024.06.026. Epub 2024 Jun 27. PMID 38937182